CLINICAL TRIAL: NCT03111719
Title: Human Brown Adipose Tissue Histological and Mitochondrial Respiratory Analysis
Brief Title: Human Brown Adipose Tissue and Mitochondrial Respiration
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Ministry of Education, Culture and Science (Unknown)
Responsible Party: Sponsor
Other Study IDs: NL31367.068.10
Record Dates: First submitted 2017-03-30; First posted 2017-04-13 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Mitochondrial Metabolism Disorders; Adipose Tissue, Brown; Aging; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
This study is focused on measuring mitochondrial activity of human brown adipose tissue. During surgery, adipose tissue biopsies from white and brown adipose tissue will be collected from the deep neck area. These biopsies will be used to examine mitochondrial function via histological analysis, biochemical analysis and in vitro experiments based on precursor cells present in the biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Indication for surgery in the supraclavicular and neck region (more specific patients diagnosed with hyperparathyroidism, struma, benign thyroid gland tumours, implantation of a vagal neurostimulator for epilepsia and cervical neurologic disorders)
* In the thyroid gland group, euthyroid function

Exclusion Criteria:

* Pre-operatively diagnosed malign tumour
* Patients undergoing acute surgery because of critical illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated for surgery in the supraclavicular and neck region
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2010-01-04 (Actual); Primary Completion 2021-10-10 (Estimated); Study Completion 2021-10-10 (Estimated)

PRIMARY OUTCOMES:
Mitochondrial respiration in human brown | 8 weeks
  Measure of mitochondrial respiration in human brown adipose tissue biopsies and measure mitochondrial respiration in cells derived from human brown adipose tissue biopsies. With high resolution respirometry , oxygen consumption in mitochondria will be determined using different substrates that stimulate mitochondrial activity including norepinephrine which is a natural agonist to increase mitochondrial activity in brown adipose tissue. During these experiments mitochondrial complex activity can be inhibited using specific inhibitors.

SECONDARY OUTCOMES:
Characterise human brown adipose tissue | 8 weeks
  Perform histological analysis and biochemical analysis in brown adipose tissue biopsies and compare to skeletal muscle. Via qPCR analysis, western blotting and immunfluorescence we will examine UCP1 expression in BAT.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center / University of Maastricht, Maastricht, Netherlands

REFERENCES:
- [Derived] Nascimento EBM, Moonen MPB, Remie CME, Gariani K, Jorgensen JA, Schaart G, Hoeks J, Auwerx J, van Marken Lichtenbelt WD, Schrauwen P. Nicotinamide Riboside Enhances In Vitro Beta-adrenergic Brown Adipose Tissue Activity in Humans. J Clin Endocrinol Metab. 2021 Apr 23;106(5):1437-1447. doi: 10.1210/clinem/dgaa960. PMID 33524145
- [Derived] Nascimento EBM, Sparks LM, Divoux A, van Gisbergen MW, Broeders EPM, Jorgensen JA, Schaart G, Bouvy ND, van Marken Lichtenbelt WD, Schrauwen P. Genetic Markers of Brown Adipose Tissue Identity and In Vitro Brown Adipose Tissue Activity in Humans. Obesity (Silver Spring). 2018 Jan;26(1):135-140. doi: 10.1002/oby.22062. Epub 2017 Nov 27. PMID 29178600